CLINICAL TRIAL: NCT02349542
Title: The Safety of Liposomal Bupivacaine in Simultaneous Bilateral Total Knee Arthroplasty
Brief Title: Liposomal Bupivacaine in Simultaneous Bilateral Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-14-10B
Record Dates: First submitted 2015-01-16; First posted 2015-01-29 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Arthroplasty, Replacement, Knee; Pain
Keywords: Liposomal Bupivacaine; Simultaneous Bilateral Total Knee Arthroplasty; Safety
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liposomal bupivacaine (Experimental): Patients will receive liposomal bupivacaine following simultaneous bilateral total knee arthroplasty.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — One (1) 20 mL vial of 266 mg liposomal bupivacaine (3% (~8mg free bupivacaine)) will be injected into each surgical (knee) site following simultaneous bilateral total knee arthroplasty. In addition, 30 mL of 0.25% bupivacaine (75 mg free bupivacaine) will be injected into each surgical (knee) site for a total of 83 mg free bupivacaine injected into each surgical (knee) site.
  Other Names: Exparel

SUMMARY:
The purpose of this study is to evaluate the serum levels (pharmacokinetics) of bupivacaine in a series of patients undergoing simultaneous bilateral total knee arthroplasty with the use of a standardized periarticular injection containing free bupivacaine and liposomal bupivacaine.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a commonly performed and successful surgical procedure that has been shown to dramatically decrease pain and improve patient's function and quality of life. Certain patients may present with significant pain and limitations due to pain in both knees and based on age, health and degree of deformity may be candidates for bilateral simultaneous total knee arthroplasty. The safety and efficacy of simultaneous bilateral total knee arthroplasty has been well documented in the literature.

Inadequate postoperative pain control following TKA has been one of the greatest sources of patient dissatisfaction following total knee arthroplasty. Traditionally, it has been managed with parenteral and oral narcotics. Recently, a number of studies have demonstrated the efficacy of multimodal analgesia following a variety of surgical procedures. These multimodal regimens vary and consist of any number of medications including non-steroidal anti-inflammatories, anti-epileptics, and peripheral nerve blocks among others. These multimodal regimens have been associated with a reduction in the use of opioid analgesics, leading to fewer opioid-associated adverse events.

One of the newest modalities introduced on the market is liposomal bupivacaine (Exparel). Liposomal bupivacaine is a lipid encapsulated bupivacaine that allows for depo administration of the medication into the soft tissue during a surgical procedure. The lipids are engineered to slowly release over an approximately 72 hour time period, resulting in the slow release of free bupivacaine in to the soft tissue of the surgical site. This has the proposed advantage of a longer duration of analgesia compared to standard bupivacaine injections.

Liposomal bupivacaine is applied in a periarticular injection at the conclusion of TKAs to aid in post-operative pain control. Due to the lipid encapsulation of the bupivacaine, only 3% free bupivacaine is released into the tissue at initial infiltration, with the remainder released slowly over approximately a 72 hour time frame. To cover, this gap period, the liposomal bupivacaine is mixed with standard bupivacaine to allow for an immediate analgesic effect.

A potential risk, although low, is the concern for bupivacaine toxicity. Toxicity from bupivacaine is associated with central nervous system issues (seizures) and cardiac toxicity. Toxicity is dose dependent and recommended levels should not exceed 400mg/24 hr period. With the use of bupivacaine into each surgical site, there is a theoretical risk, if administered intra-vascularly, of bupivacaine toxicity. To date, no study has evaluated the safety of liposomal bupivacaine when used in simultaneous bilateral total knee arthroplasty. The use of liposomal bupivacaine is FDA approved for infiltration of one vial into one surgical site. Other specialties have evaluated the use of one vial of liposomal bupivacaine into two surgical sites (breast augmentation) at one surgery without any adverse events.

To date, approximately 8-10 patients at the investigator's institution have undergone simultaneous bilateral total knee arthroplasty with the use of liposomal bupivacaine without a known adverse event. A recent study published by Bramlett (2012) used 2 vials (532mg) in one knee to evaluate efficacy. There were no changes in patient's vitals signs or cardiac events in those patients receiving liposomal bupivacaine at the highest dose. In addition, a study by Bergese looked at doses of up to 600mg of liposomal bupivacaine in a Phase 2 safety study and found no adverse cardiac events. The purpose of this study is to evaluate the serum levels (pharmacokinetics) of bupivacaine in a series of patients undergoing simultaneous bilateral total knee arthroplasty with the use of a standardize periarticular injection containing free bupivacaine and liposomal bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed appropriate candidates for simultaneous bilateral total knee arthroplasty.
* Patients receiving general anesthesia
* Understands the local language and is willing and able to follow the requirements of the protocol
* Understands the informed consent and signs the institutional review board/ independent ethics committee (IRB/IEC) approved informed consent form

Exclusion Criteria:

* Patients less than 18 years of age
* Allergy to bupivacaine
* Allergy to epinephrine
* Patients who are not medically cleared to undergo bilateral total knee replacement surgery, or
* Patient-reported liver impairment (per investigator discretion)
* Patient-reported renal impairment (per investigator discretion)
* Patients receiving spinal anesthesia
* Females who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Odum, PhD, Study Director — Senior Research Scientist; Bryan D Springer, MD, Principal Investigator — Physician
Locations (1):
- OrthoCarolina, PA, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Bosco JA 3rd, Slover JD, Haas JP. Perioperative strategies for decreasing infection: a comprehensive evidence-based approach. J Bone Joint Surg Am. 2010 Jan;92(1):232-9. No abstract available. PMID 20048118
- [Background] Zeni JA Jr, Snyder-Mackler L. Clinical outcomes after simultaneous bilateral total knee arthroplasty: comparison to unilateral total knee arthroplasty and healthy controls. J Arthroplasty. 2010 Jun;25(4):541-6. doi: 10.1016/j.arth.2009.02.016. Epub 2009 Apr 7. PMID 19356894
- [Background] Taylor BC, Dimitris C, Mowbray JG, Gaines ST, Steensen RN. Perioperative safety of two-team simultaneous bilateral total knee arthroplasty in the obese patient. J Orthop Surg Res. 2010 Jun 17;5:38. doi: 10.1186/1749-799X-5-38. PMID 20565781
- [Background] Shin YH, Kim MH, Ko JS, Park JA. The safety of simultaneous bilateral versus unilateral total knee arthroplasty: the experience in a Korean hospital. Singapore Med J. 2010 Jan;51(1):44-9. PMID 20200775
- [Background] Kim SY, An YJ, Kim SH, Kim HK, Park JS, Shin YS. The effect of postoperative pain on postoperative blood loss after sequential bilateral total knee arthroplasty. Korean J Anesthesiol. 2011 Feb;60(2):98-102. doi: 10.4097/kjae.2011.60.2.98. Epub 2011 Feb 25. PMID 21390164
- [Background] Parvizi J, Miller AG, Gandhi K. Multimodal pain management after total joint arthroplasty. J Bone Joint Surg Am. 2011 Jun 1;93(11):1075-84. doi: 10.2106/JBJS.J.01095. PMID 21655901
- [Background] Goyal N, McKenzie J, Sharkey PF, Parvizi J, Hozack WJ, Austin MS. The 2012 Chitranjan Ranawat award: intraarticular analgesia after TKA reduces pain: a randomized, double-blinded, placebo-controlled, prospective study. Clin Orthop Relat Res. 2013 Jan;471(1):64-75. doi: 10.1007/s11999-012-2596-9. PMID 23011843
- [Background] Hutchinson RW, Chon EH, Gilder R, Moss J, Daniel P. A comparison of a fentanyl, morphine, and hydromorphone patient-controlled intravenous delivery for acute postoperative analgesia: a multicenter study of opioid-induced adverse reactions. Hospital Pharmacy 41(7): 659-663, 2006.
- [Background] Jin F, Chung F. Multimodal analgesia for postoperative pain control. J Clin Anesth. 2001 Nov;13(7):524-39. doi: 10.1016/s0952-8180(01)00320-8. PMID 11704453
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Horlocker TT, Hebl JR, Kinney MA, Cabanela ME. Opioid-free analgesia following total knee arthroplasty--a multimodal approach using continuous lumbar plexus (psoas compartment) block, acetaminophen, and ketorolac. Reg Anesth Pain Med. 2002 Jan-Feb;27(1):105-8. doi: 10.1053/rapm.2002.27177. PMID 11799514
- [Background] Lombardi AV Jr, Berend KR, Mallory TH, Dodds KL, Adams JB. Soft tissue and intra-articular injection of bupivacaine, epinephrine, and morphine has a beneficial effect after total knee arthroplasty. Clin Orthop Relat Res. 2004 Nov;(428):125-30. doi: 10.1097/01.blo.0000147701.24029.cc. PMID 15534532
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Minkowitz HS, Onel E, Patronella CK, Smoot JD. A two-year observational study assessing the safety of DepoFoam bupivacaine after augmentation mammaplasty. Aesthet Surg J. 2012 Feb;32(2):186-93. doi: 10.1177/1090820X11434524. Epub 2012 Jan 11. PMID 22238339

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine
Started | 20
Completed (Patients were withdrawn from the study if they did not schedule surgery or canceled their surgery.) | 15
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Liposomal Bupivacaine
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 60 [57 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Body Mass Index [Mean (Full Range); unit: kilograms per meters-squared] | 30.7 [27 to 34.9]

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of Participants with Adverse Events
Time Frame: Up to 72 hours following injection
Measure: Number; unit: participants
Arm/Group | Liposomal Bupivacaine
Number analyzed (Participants) | 15
participants | 0

2. Secondary Outcome: Plasma Bupivacaine Levels
Description: Blood samples will be drawn and analyzed to establish levels of bupivacaine detectable in the blood. Blood samples will be drawn at baseline (prior to injection), upon injection, at 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours post-injection and analyzed to determine levels of bupivacaine present.
Time Frame: Up to 72 hours following injection
Population: Blood draws were collected at the pre-defined intervals unless the patient was discharged prior to the blood collection time. 6 patients were discharged prior to the 48 hour collection time. 5 additional patients were discharged prior to the 72 hour collection time.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Liposomal Bupivacaine
Number analyzed (Participants) | 15
ug/ml
  Baseline (Pre-Injection) | 0 (0)
  Immediately Following Injection | 0.22 (0.25)
  15 minutes after injection | 0.31 (0.25)
  30 minutes after injection | 0.35 (0.21)
  1 hour after injection | 0.47 (0.21)
  2 hours after injection | 0.53 (0.21)
  4 hours after injection | 0.56 (0.26)
  8 hours after injection | 0.63 (0.20)
  12 hours after injection | 0.56 (0.25)
  24 hours after injection | 0.71 (0.22)
  48 hours after injection: number analyzed (Participants) | 9
  48 hours after injection | 0.80 (0.37)
  72 hours after injection: number analyzed (Participants) | 4
  72 hours after injection | 0.43 (0.22)

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events through the 6-week follow-up visit.
Arm/Group | Liposomal Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No